CLINICAL TRIAL: NCT02898571
Title: Cross-over Double-blind Intervention to Investigate the Effects of Defined Antioxidant-containing Drinks on Time Course of Antioxidant Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anthony Watson, NU-Food Facility Manager, Newcastle University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NUHEALTH-KB002-AC
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: The Impact of Vitamin c and Epicatechin Upon Antioxidant Capactity
MeSH Terms: interventions — Ascorbic Acid; Catechin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 360ml water based drink containing 50g mix of glucose and fructose plus flavouring
  Interventions: Dietary Supplement: Placebo
- Vitamin C (Experimental): 360ml water based drink containig 60mg vitamin C and 50g mix of glucose and fructose plus flavouring
  Interventions: Dietary Supplement: Vitamin C
- Epicatechin (Experimental): 360ml water based drink containig 80mg epicatechin and 50g mix of glucose and fructose plus flavouring
  Interventions: Dietary Supplement: epicatechin

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo comparitor
  Arms: Placebo
Dietary Supplement: Vitamin C — Active treatment
  Arms: Vitamin C
Dietary Supplement: epicatechin — Active treatment
  Arms: Epicatechin

SUMMARY:
The aim of this project is to measure the differences in antioxidant capacity at different time points after consuming a single dose of antioxidant-containing drink (vitamin C or epicatechin) compared with a control drink in 10 volunteers, and then match the data with the proposed modelling corresponding to either homeostasis or accumulation. Additionally it will also determine whether the effect on changes of antioxidant capacity in response to epicatechin and vitamin c is equal.

DETAILED DESCRIPTION:
The sample size is 10 volunteers. This was based on an estimate of the number of datasets required to ensure that at least some of the datasets show time courses that are suitable for the demonstration. The trial uses a cross-over double-blind placebo-controlled design.

A participant information sheet will be given to the participant to read at least 24 hours prior to the screening. Eligibility of participants will be checked during the screening session. The participant anthropometric measurements (height, weight, body fat) will be taken and a Health Questionnaire will be filled completed.

Inclusion Criteria: Healthy adults, BMI 18.5-30

Exclusion Criteria: Any disease or medication that affects metabolism or digestion, smokers, common cold or other inflammatory illness at the time of bio-sample collection. Any other physical or mental condition that in the judgement of the experimenter would mean that participation in the study would be an undue burden on the volunteer.

At the screening session, the participant will be informed the relevant details of the study. Specifically they must avoid consumption of fruits, vegetables and whole grain products, coffee and tea, beer and wine for 48 hours before the start of the intervention and 24 hours after it (however cola, 7-up and similar caffeine-containing drinks without any real fruits or herbs are fine). After they have had opportunity to ask any questions regarding the testing procedures, if they are happy to take part, they will be free to ask and sign a consent form.

Antioxidant Intervention Session:

Overall, each volunteer will be randomised to receive three treatments in a crossover design, one with epicatechin containing drink as treatment, one with vitamin C and another without antioxidants as placebo.

The volunteers will avoid consumption of fruits, vegetables and whole grain products, coffee and tea, beer and wine for 48 hours before the intervention and 24 hours after it, and the intervention will be administered after an overnight fast (12 hours). At each test, the volunteer will consume 360ml of drink, with either 60mg vitamin C corresponding to a smoothie, or 80 mg epicatechin corresponding to approx. 56g unsweetened baking chocolate (Bhagwat, 2014) or no antioxidant (placebo) and all containing 13% sugar (providing 50g a mixture of glucose and fructose) and a relevant flavouring.

The optimal timing of samples has been determined using mathematical models of the results from the initial study done for BBC with the help of Professor Gunnar Cedersund (Linköping University). Capillary blood samples will be obtained by finger prick and collected in multivette 600 tubes (600µl per tube). at baseline, 0, 0.5, 1, 1.5, 2, 2.5, 3.5, 5, 6, 8 and 24 hours post dose. Breakfast will be served between 1.5 and 2 hours after consumption of the drink, and lunch after the 3.5-hour sample has been collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults,
* BMI 18.5-30

Exclusion Criteria:

* Any disease or medication that affects metabolism or digestion, smokers, common cold or other inflammatory illness at the time of bio-sample collection. Any other physical or mental condition that in the judgement of the experimenter would mean that participation in the study would be an undue burden on the volunteer

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Antioxidant capacity | Baseline 0, 0.5, 1, 1.5, 2, 2.5, 3.5, 5, 6, 8 and 24 hours post dose
  measure the differences in antioxidant capacity at different time point after consuming a single dose of antioxidant-containing drink (vitamin C or epicatechin) compared with a control and then match the data with the proposed modelling corresponding to either homoeostasis or accumulation.

SECONDARY OUTCOMES:
Antioxidant capacity of epicatechin and vitamin-C | Baseline 0, 0.5, 1, 1.5, 2, 2.5, 3.5, 5, 6, 8 and 24 hours post dose
  etermine whether the effect on changes of antioxidant capacity in response to epicatechin and vitamin c is equal

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom